CLINICAL TRIAL: NCT03153137
Title: Prospective, Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study Assessing the Efficacy and Safety of Macitentan in Fontan-palliated Adult and Adolescent Subjects
Brief Title: Clinical Study Assessing the Efficacy and Safety of Macitentan in Fontan-palliated Subjects
Acronym: RUBATO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-055H301; 2016-003320-23 (EudraCT Number)
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Macitentan (Experimental): Macitentan 10 mg per day; film-coated tablet; oral use
  Interventions: Drug: Macitentan 10 mg
- Placebo (Placebo Comparator): film-coated tablet; oral use
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Macitentan 10 mg — film-coated tablet; oral use
  Arms: Macitentan
Drug: Placebo — film-coated tablet; oral use
  Arms: Placebo

SUMMARY:
The primary objective is to assess the effect of macitentan 10 mg as compared to placebo on exercise capacity through cardiopulmonary exercise testing.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent from the subject and/or a legal representative prior to initiation of any study-mandated procedures
* Fontan-palliated subjects with either intra-atrial lateral tunnel total cavopulmonary connection (LT-TCPC), or extra cardiac tunnel TCPC (EC-TCPC) surgery > 1 year before Screening. Either LT- or EC-TCPC can be primary or secondary to atrio-pulmonary connection
* New York Heart Association (NYHA) functional class (FC) II or III (assessed by the investigator using the Specific Activity Scale
* Women of childbearing potential must have a negative serum pregnancy test use reliable contraception

Exclusion Criteria:

* Pattern of Fontan circulation severity
* Deterioration of the Fontan-palliated condition.
* Limitations to Cardiopulmonary exercise testing (CPET)
* Peak VO2 < 15 mL/kg/min.
* Any known factor or disease that may interfere with treatment compliance or full participation in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - Massachusetts General Hospital Heart Center, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Providence Medical Research Providence Health Care, Spokane, Washington
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Camperdown
  - The Prince Charles Hospital, Adult Congenital Heart Disease Unit, Chermside
  - Royal Children's Hospital, Parkville
  - Queensland CHILDREN'S HOSPITAL, South Brisbane
  - Westmead Hospital, Westmead
- CHU de Quebec Universite Laval, Québec, Quebec, Canada
- China (4):
  - Beijing Anzhen Hospital, Beijing
  - Beijing Fuwai Hospital, Beijing
  - Shanghai Childrens Medical Center, Shanghai
  - Wuhan Asia Heart Hospital, Wuhan
- Fakultni nemocnice v Motole, Prague, Czechia
- Rigshospitalet Kardiologisk Klinisk, Copenhagen, Denmark
- France (3):
  - CHU Arnaud de Villeneuve, Montpellier
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital Cardiologique Du Haut-Lévêque, Pessac
- Germany (2):
  - Deutsches Herzzentrum Berlinklinik Für Angeborene Herzfehler, Berlin
  - Deutsches Herzzentrum München, München
- Auckland City Hospital, Auckland, New Zealand
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Krakowski Szpital Specjalityczny im Jana Pawla II Oddzial Kliniczny Chorob Serca i Naczyn, Krakow
  - Wojewodzki Szpital Specjalistyczny We Wroclawiu, Wroclaw
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - Birmingham Children's Hospital, Birmingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 142 participants were enrolled, out of which 137 participants were included in the analysis as 5 participants were excluded due to regulatory restrictions.
Groups:
- Placebo: Participants received Macitentan matching placebo tablet orally, once daily with or without food starting at Week 0 up to Week 52.
- Macitentan: Participants received Macitentan 10 milligrams (mg) tablet, orally once daily with or without food starting at Week 0 up to Week 52.
Period: Overall Study
Arm/Group | Placebo | Macitentan
Started | 69 | 68
Completed | 66 | 64
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Macitentan | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (7.49) | 23.2 (5.82) | 23.9 (6.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 44 | 45 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 59 | 58 | 117
  Unknown or Not Reported | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 52 | 55 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 7 | 7 | 14
  Canada | 1 | 3 | 4
  China | 3 | 3 | 6
  Czech Republic | 9 | 11 | 20
  Denmark | 10 | 13 | 23
  France | 5 | 4 | 9
  New Zealand | 1 | 2 | 3
  Poland | 17 | 9 | 26
  Taiwan, Province Of China | 4 | 2 | 6
  United Kingdom | 1 | 3 | 4
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Oxygen Uptake/Consumption (VO2) Up to Week 16
Description: Change from baseline in peak VO2 up to Week 16 was reported.
Time Frame: Baseline up to Week 16
Population: Full analysis set (FAS) included all participants randomized to the study treatment.
Measure: Mean (Standard Deviation); unit: Milliliter/kilogram/minute (mL/kg/min)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
Milliliter/kilogram/minute (mL/kg/min) | -0.67 (2.657) [lower limit 2.657] | -0.16 (2.855) [lower limit 2.855]
Statistical Analysis 1: Comparison: Placebo vs Macitentan; Due to adaptive nature of the design, the main analysis was conducted on FAS using the inverse normal combination method with pre-specified weights to combine first and second stage p-values; Test type: Superiority — For each stage, the p-value from the ANCOVA model including randomized treatment, geographical region, and baseline peak VO2 was used to construct the final adjusted p-value; p = 0.1930, ANCOVA — Final adjusted p-value (from weighted inverse normal combination test); Median unbiased estimate and repeated CI = 0.62, 99% CI 2-sided [-0.62 to 1.85]

2. Secondary Outcome: Change From Baseline in Peak VO2 Up to Week 52
Description: Change from baseline in peak VO2 up to Week 52 was reported.
Time Frame: Baseline up to Week 52
Population: FAS included all participants randomized to the study treatment.
Measure: Least Squares Mean (Standard Error); unit: mL/kg/min
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
mL/kg/min | -0.92 (0.296) [lower limit 0.296] | -0.31 (0.293) [lower limit 0.293]

3. Secondary Outcome: Change From Baseline in Mean Count Per Minute of Daily Physical Activity Measured by Accelerometer (PA-Ac) Up to Week 16
Description: Change from baseline in mean count per minute of daily PA-Ac up to Week 16 was reported. The daily physical activity (counts per min) of the participant was assessed via accelerometer during daytime. The accelerometer was given to the participant at Visit 1, and data was collected for 9 consecutive daily daytime periods after Visit 1 (baseline) to Visit 4 (Week 16).
Time Frame: Baseline up to Week 16
Population: FAS included all participants randomized to the study treatment. Here, N (number of participants analyzed) is defined as the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: counts per minute
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 58 | 61
counts per minute | -14.34 (117.562) | -3.02 (92.443)

4. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 56 weeks
Population: The Safety analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
Participants | 9 | 13

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 56 weeks
Population: The Safety analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
Participants | 44 | 48

6. Secondary Outcome: Number of Participants With AEs Leading to Premature Discontinuation of Study Treatment
Description: Number of participants with AEs leading to premature discontinuation of study treatment was reported. AEs leading to premature discontinuation of study treatment were those with action taken with study drug reported as 'permanently discontinued' by the investigator.
Time Frame: Up to 56 weeks
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
Participants | 1 | 3

7. Secondary Outcome: Change From Baseline in Systolic and Diastolic Arterial Blood Pressure (BP)
Description: Change from baseline in systolic and diastolic arterial BP at Week 8, Week 16, Week 32 and Week 52 was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: Safety analysis set included all participants who received at least one dose of study treatment. Here, N (number of participants analyzed) signifies participants evaluable for this outcome measure. Here "n" signifies number of participants evaluable at different timepoints.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
millimeters of mercury (mmHg)
  Baseline | 116.0 (12.10) | 117.0 (10.95)
  Systolic BP: Week 8: number analyzed (Participants) | 33 | 38
  Systolic BP: Week 8 | 2.5 (14.41) | -0.4 (11.67)
  Systolic BP: Week 16: number analyzed (Participants) | 66 | 65
  Systolic BP: Week 16 | 0.5 (14.68) | -4.6 (13.05)
  Systolic BP: Week 32: number analyzed (Participants) | 17 | 24
  Systolic BP: Week 32 | -6.3 (15.09) | -3.1 (10.51)
  Systolic BP: Week 52: number analyzed (Participants) | 60 | 59
  Systolic BP: Week 52 | 0.0 (12.12) | -4.8 (12.08)
  Diastolic BP: Week 8: number analyzed (Participants) | 33 | 38
  Diastolic BP: Week 8 | -0.2 (5.86) | -0.1 (9.57)
  Diastolic BP: Week 16: number analyzed (Participants) | 66 | 65
  Diastolic BP: Week 16 | -0.6 (10.06) | -3.1 (8.74)
  Diastolic BP: Week 32: number analyzed (Participants) | 17 | 24
  Diastolic BP: Week 32 | 1.3 (8.64) | -1.4 (8.21)
  Diastolic BP: Week 52: number analyzed (Participants) | 60 | 59
  Diastolic BP: Week 52 | 1.3 (10.84) | -2.8 (11.21)

8. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change from baseline in pulse rate at Week 8, Week 16, Week 32 and Week 52 was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: Safety analysis set included all participants who received at least one dose of study treatment. Here "n" signifies number of participants evaluable at different timepoints.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
beats per minute (bpm)
  Baseline | 81.3 (12.52) | 78.2 (13.33)
  Week 8: number analyzed (Participants) | 33 | 38
  Week 8 | -3.9 (12.80) | -5.9 (12.07)
  Week 16: number analyzed (Participants) | 66 | 65
  Week 16 | 0.1 (14.76) | -0.1 (11.57)
  Week 32: number analyzed (Participants) | 17 | 24
  Week 32 | 0.2 (12.37) | 1.1 (9.10)
  Week 52: number analyzed (Participants) | 60 | 59
  Week 52 | -0.7 (11.56) | -2.9 (10.25)

9. Secondary Outcome: Change From Baseline in Oxygen Saturation (SpO2)
Description: Change from baseline in SpO2 was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: Safety set included all participants who received at least one dose of study treatment. Here "n" signifies number of participants evaluable at different timepoints.
Measure: Mean (Standard Deviation); unit: percent of oxygen saturation
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
percent of oxygen saturation
  Baseline | 92.6 (3.22) | 92.8 (2.84)
  Week 8: number analyzed (Participants) | 32 | 37
  Week 8 | 0.0 (3.20) | 1.2 (2.78)
  Week 16: number analyzed (Participants) | 66 | 65
  Week 16 | 0.5 (2.57) | 0.8 (2.75)
  Week 32: number analyzed (Participants) | 17 | 23
  Week 32 | 0.8 (2.94) | 1.4 (3.73)
  Week 52: number analyzed (Participants) | 60 | 59
  Week 52 | 1.4 (2.77) | 0.9 (2.99)

10. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
kilograms (kg)
  Baseline | 68.89 (17.296) | 67.38 (14.721)
  Week 8: number analyzed (Participants) | 33 | 38
  Week 8 | -0.38 (1.996) | 0.43 (1.568)
  Week 16: number analyzed (Participants) | 66 | 65
  Week 16 | 0.21 (2.028) | 0.58 (2.230)
  Week 32: number analyzed (Participants) | 19 | 27
  Week 32 | 0.73 (2.952) | 0.77 (3.411)
  Week 52: number analyzed (Participants) | 60 | 59
  Week 52 | 1.44 (3.746) | 1.30 (4.358)

11. Secondary Outcome: Number of Participants With Treatment-emergent Markedly Abnormal Laboratory Values
Description: Number of participants with treatment-emergent markedly laboratory abnormal laboratory values were reported. Abnormal values for platelets (LL < 75); Lymphocytes (HH > 4.0); Neutrophils (LL < 1.5); Prothrombin International Normalized Ratio: HH (greater than and equal to [>=] 1.5 upper limit of normal [ULN]), Ratio: HH >= 2.5 ULN); Bilirubin (HH >= 2 ULN); Alkaline Phosphatase (HH > 2.5 ULN); Glomerular Filtration Rate (LL < 60); Glucose (HH > 8.9); Triglycerides (HH > 3.42). Here "HH" refers to values above the normal range, where H stands for "high" and "LL" refers to values below the normal range where L stands for "low".
Time Frame: Up to 56 weeks
Population: Safety analysis set included all participants who received at least one dose of study treatment. Here, N (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 67
Participants
  Platelets: LL (< 75) | 2 | 1
  Lymphocytes: HH (> 4.0) | 0 | 1
  Neutrophils: LL (< 1.5) | 0 | 2
  Prothrombin International Normalized Ratio: HH (>= 1.5 ULN) | 3 | 5
  Prothrombin International Normalized Ratio: HH (>= 2.5 ULN) | 1 | 1
  Bilirubin: HH (>= 2 ULN) | 1 | 2
  Alkaline Phosphatase: HH (> 2.5 ULN) | 1 | 0
  Glomerular Filtration Rate: LL (< 60): number analyzed (Participants) | 68 | 67
  Glomerular Filtration Rate: LL (< 60) | 1 | 1
  Glucose: LL (< 3.0): number analyzed (Participants) | 68 | 67
  Glucose: LL (< 3.0) | 0 | 2
  Glucose: HH (> 8.9): number analyzed (Participants) | 68 | 67
  Glucose: HH (> 8.9) | 0 | 2
  Triglycerides: HH (> 3.42): number analyzed (Participants) | 68 | 67
  Triglycerides: HH (> 3.42) | 3 | 1

12. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Change from baseline in hemoglobin was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: Safety analysis set included all participants who received at least one dose of study treatment. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here "n" signifies number of participants evaluable at different timepoints.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 67
grams per liter (g/L)
  Baseline | 160.4 (13.43) | 159.5 (12.83)
  Week 8: number analyzed (Participants) | 57 | 58
  Week 8 | 0.0 (6.59) | -8.7 (9.33)
  Week 16: number analyzed (Participants) | 62 | 64
  Week 16 | 0.0 (7.75) | -8.7 (8.51)
  Week 32: number analyzed (Participants) | 52 | 51
  Week 32 | 1.3 (8.29) | -7.3 (9.84)
  Week 52: number analyzed (Participants) | 59 | 55
  Week 52 | -2.9 (10.04) | -7.1 (10.02)

13. Secondary Outcome: Change From Baseline in Hematocrit
Description: Change from baseline in hematocrit was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liter/Liter (L/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 67
Liter/Liter (L/L)
  Baseline | 0.472 (0.041) | 0.471 (0.034)
  Week 8: number analyzed (Participants) | 35 | 38
  Week 8 | 0.002 (0.027) | -0.030 (0.023)
  Week 16: number analyzed (Participants) | 62 | 63
  Week 16 | 0.003 (0.027) | -0.023 (0.026)
  Week 32: number analyzed (Participants) | 19 | 24
  Week 32 | 0.003 (0.031) | -0.009 (0.028)
  Week 52: number analyzed (Participants) | 59 | 55
  Week 52 | -0.010 (0.030) | -0.021 (0.028)

14. Secondary Outcome: Change From Baseline in Erythrocytes and Reticulocytes
Description: Change from baseline in erythrocytes and reticulocytes at Week 8, Week 16, Week 32 and Week 52 was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 68 | 64
10^12 cells per liter
  Erythrocytes: Baseline: number analyzed (Participants) | 65 | 63
  Erythrocytes: Baseline | 5.251 (0.4832) | 5.205 (0.3544)
  Erythrocytes: Week 8: number analyzed (Participants) | 31 | 34
  Erythrocytes: Week 8 | 0.048 (0.2461) | -0.297 (0.2866)
  Erythrocytes: Week 16: number analyzed (Participants) | 58 | 59
  Erythrocytes: Week 16 | 0.012 (0.2521) | -0.264 (0.2790)
  Erythrocytes: Week 32: number analyzed (Participants) | 16 | 20
  Erythrocytes: Week 32 | -0.031 (0.2442) | -0.090 (0.2337)
  Erythrocytes: Week 52: number analyzed (Participants) | 56 | 51
  Erythrocytes: Week 52 | -0.096 (0.2515) | -0.184 (0.2671)
  Reticulocytes: Baseline: | 0.075 (0.028) | 0.070 (0.022)
  Reticulocytes: Week 8: number analyzed (Participants) | 33 | 32
  Reticulocytes: Week 8 | -0.006 (0.017) | -0.006 (0.016)
  Reticulocytes: Week 16: number analyzed (Participants) | 61 | 60
  Reticulocytes: Week 16 | -0.003 (0.026) | -0.001 (0.021)
  Reticulocytes: Week 32: number analyzed (Participants) | 18 | 19
  Reticulocytes: Week 32 | -0.003 (0.028) | -0.008 (0.027)

15. Secondary Outcome: Change From Baseline in Leucocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils and Platelets
Description: Change from baseline in leucocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelets at Week 8, Week 16, Week 32 and Week 52 was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 67
10^9 cells per liter
  Leukocytes: Baseline | 6.270 (1.7553) | 5.693 (1.5679)
  Leukocytes: Week 8: number analyzed (Participants) | 35 | 38
  Leukocytes: Week 8 | -0.242 (1.7651) | -1.001 (1.2096)
  Leukocytes: Week 16: number analyzed (Participants) | 62 | 63
  Leukocytes: Week 16 | -0.199 (1.5490) | -0.378 (1.3908)
  Leukocytes: Week 32: number analyzed (Participants) | 19 | 24
  Leukocytes: Week 32 | 0.417 (1.1782) | -0.237 (1.7224)
  Leukocytes: Week 52: number analyzed (Participants) | 59 | 55
  Leukocytes: Week 52 | -0.554 (1.4050) | -0.715 (1.6433)
  Neutrophils: Baseline | 4.100 (1.3222) | 3.831 (1.1268)
  Neutrophils: Week 8: number analyzed (Participants) | 34 | 35
  Neutrophils: Week 8 | -0.133 (1.3604) | -0.743 (0.9864)
  Neutrophils: Week 16: number analyzed (Participants) | 62 | 63
  Neutrophils: Week 16 | -0.291 (1.3547) | -0.373 (1.0896)
  Neutrophils: Week 32: number analyzed (Participants) | 19 | 22
  Neutrophils: Week 32 | 0.494 (0.9719) | -0.254 (1.2012)
  Neutrophils: Week 52: number analyzed (Participants) | 59 | 55
  Neutrophils: Week 52 | -0.384 (1.1619) | -0.627 (1.2475)
  Lymphocytes: Baseline | 1.489 (0.6791) | 1.263 (0.4974)
  Lymphocytes: Week 8: number analyzed (Participants) | 34 | 35
  Lymphocytes: Week 8 | -0.113 (0.4770) | -0.165 (0.2886)
  Lymphocytes: Week 16: number analyzed (Participants) | 62 | 63
  Lymphocytes: Week 16 | 0.073 (0.4756) | 0.042 (0.6164)
  Lymphocytes: Week 32: number analyzed (Participants) | 19 | 22
  Lymphocytes: Week 32 | 0.047 (0.3341) | 0.126 (0.2269)
  Lymphocytes: Week 52: number analyzed (Participants) | 59 | 55
  Lymphocytes: Week 52 | -0.082 (0.4740) | -0.033 (0.3890)
  Baseline: Monocytes | 0.416 (0.1698) | 0.409 (0.1541)
  Monocytes: Week 8: number analyzed (Participants) | 34 | 35
  Monocytes: Week 8 | -0.017 (0.1645) | -0.081 (0.1400)
  Monocytes: Week 16: number analyzed (Participants) | 62 | 63
  Monocytes: Week 16 | 0.002 (0.1703) | -0.050 (0.1202)
  Monocytes: Week 32: number analyzed (Participants) | 19 | 22
  Monocytes: Week 32 | -0.018 (0.1209) | -0.071 (0.1162)
  Monocytes: Week 52: number analyzed (Participants) | 59 | 55
  Monocytes: Week 52 | -0.039 (0.1380) | -0.077 (0.1257)
  Eosinophils: Baseline | 0.207 (0.3480) | 0.151 (0.1333)
  Eosinophils: Week 8: number analyzed (Participants) | 34 | 35
  Eosinophils: Week 8 | -0.003 (0.5146) | 0.014 (0.0816)
  Eosinophils: Week 16: number analyzed (Participants) | 62 | 63
  Eosinophils: Week 16 | 0.016 (0.3056) | 0.002 (0.0755)
  Eosinophils: Week 32: number analyzed (Participants) | 19 | 22
  Eosinophils: Week 32 | -0.100 (0.5447) | 0.029 (0.1951)
  Eosinophils: Week 52: number analyzed (Participants) | 59 | 55
  Eosinophils: Week 52 | -0.046 (0.3597) | 0.015 (0.1935)
  Basophils: Baseline | 0.055 (0.0322) | 0.040 (0.0245)
  Basophils: Week 8: number analyzed (Participants) | 34 | 35
  Basophils: Week 8 | -0.002 (0.0255) | -0.002 (0.0233)
  Basophils: Week 16: number analyzed (Participants) | 62 | 63
  Basophils: Week 16 | 0.004 (0.0394) | 0.000 (0.0363)
  Basophils: Week 32: number analyzed (Participants) | 19 | 22
  Basophils: Week 32 | -0.003 (0.0354) | 0.016 (0.0313)
  Basophils: Week 52: number analyzed (Participants) | 59 | 55
  Basophils: Week 52 | -0.003 (0.0389) | 0.006 (0.0281)
  Platelets: Baseline | 184.3 (63.22) | 178.1 (54.93)
  Platelets: Week 8: number analyzed (Participants) | 35 | 37
  Platelets: Week 8 | -5.9 (32.85) | -9.1 (35.38)
  Platelets: Week 16: number analyzed (Participants) | 62 | 62
  Platelets: Week 16 | -5.4 (30.33) | -3.0 (28.77)
  Platelets: Week 32: number analyzed (Participants) | 19 | 24
  Platelets: Week 32 | -7.8 (33.46) | 8.2 (33.76)
  Platelets: Week 52: number analyzed (Participants) | 59 | 55
  Platelets: Week 52 | -11.2 (29.94) | -5.7 (31.75)

16. Secondary Outcome: Change From Baseline in Prothrombin Time
Description: Change from baseline in prothrombin time was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Seconds (sec)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 67 | 68
Seconds (sec)
  Baseline | 14.72 (7.033) | 15.37 (7.610)
  Week 8: number analyzed (Participants) | 32 | 37
  Week 8 | -0.23 (3.265) | -0.53 (4.567)
  Week 16: number analyzed (Participants) | 62 | 63
  Week 16 | 0.04 (3.921) | 0.36 (10.868)
  Week 32: number analyzed (Participants) | 17 | 21
  Week 32 | 1.45 (8.261) | 0.03 (4.135)
  Week 52: number analyzed (Participants) | 55 | 55
  Week 52 | -0.64 (3.167) | -1.20 (3.567)

17. Secondary Outcome: Change From Baseline in Prothrombin International Normalized Ratio
Description: Change from baseline in prothrombin international normalized ratio was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 67 | 68
Ratio
  Baseline | 1.434 (0.7364) | 1.516 (0.8014)
  Week 8: number analyzed (Participants) | 32 | 37
  Week 8 | -0.009 (0.3216) | -0.054 (0.4652)
  Week 16: number analyzed (Participants) | 62 | 63
  Week 16 | 0.015 (0.3806) | 0.049 (1.1653)
  Week 32: number analyzed (Participants) | 17 | 21
  Week 32 | 0.171 (0.9204) | 0.033 (0.4597)
  Week 52: number analyzed (Participants) | 55 | 55
  Week 52 | -0.044 (0.3265) | -0.120 (0.3889)

18. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Alkaline Phosphatase (AP)
Description: Change from baseline in ALT, AST and AP were reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
Units per liter (U/L)
  ALT: Baseline | 26.7 (9.47) | 28.5 (12.84)
  ALT: Week 8: number analyzed (Participants) | 57 | 60
  ALT: Week 8 | -0.8 (5.57) | -1.8 (9.99)
  ALT: Week 16: number analyzed (Participants) | 63 | 64
  ALT: Week 16 | -0.2 (6.86) | -1.6 (7.94)
  ALT: Week 32: number analyzed (Participants) | 52 | 51
  ALT: Week 32 | -0.4 (5.62) | -2.1 (12.53)
  ALT: Week 52: number analyzed (Participants) | 58 | 57
  ALT: Week 52 | -0.2 (8.11) | -0.3 (14.04)
  AST: Baseline | 25.8 (7.40) | 28.3 (20.95)
  AST: Week 8: number analyzed (Participants) | 56 | 59
  AST: Week 8 | -0.7 (4.92) | -4.4 (2.37)
  AST: Week 16: number analyzed (Participants) | 62 | 64
  AST: Week 16 | -0.5 (6.13) | -3.9 (20.25)
  AST: Week 32: number analyzed (Participants) | 51 | 50
  AST: Week 32 | 0.9 (4.14) | -4.7 (22.46)
  AST: Week 52: number analyzed (Participants) | 58 | 58
  AST: Week 52 | -0.6 (6.83) | -3.2 (24.16)
  AP: Baseline | 106.4 (83.54) | 100.2 (88.62)
  AP: Week 8: number analyzed (Participants) | 34 | 37
  AP: Week 8 | -7.6 (19.82) | -8.5 (18.14)
  AP: Week 16: number analyzed (Participants) | 64 | 63
  AP: Week 16 | -4.7 (19.20) | -7.1 (22.54)
  AP: Week 32: number analyzed (Participants) | 19 | 24
  AP: Week 32 | -10.1 (32.43) | -1.1 (26.30)
  AP: Week 52: number analyzed (Participants) | 59 | 57
  AP: Week 52 | -12.9 (34.81) | -7.0 (27.63)

19. Secondary Outcome: Change From Baseline in Bilirubin and Direct Bilirubin
Description: Change from baseline in bilirubin and direct bilirubin was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micromole per liter (umol/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
micromole per liter (umol/L)
  Bilirubin: Baseline | 14.65 (5.815) | 17.28 (13.379)
  Bilirubin: Week 8: number analyzed (Participants) | 34 | 37
  Bilirubin: Week 8 | 0.62 (5.985) | -1.08 (5.693)
  Bilirubin: Week 16: number analyzed (Participants) | 62 | 63
  Bilirubin: Week 16 | 1.98 (5.799) | -1.76 (7.075)
  Bilirubin: Week 32: number analyzed (Participants) | 19 | 24
  Bilirubin: Week 32 | 1.47 (5.285) | 0.29 (5.052)
  Bilirubin: Week 52: number analyzed (Participants) | 59 | 58
  Bilirubin: Week 52 | 0.69 (5.778) | -1.02 (5.778)
  Direct Bilirubin: Baseline: number analyzed (Participants) | 67 | 68
  Direct Bilirubin: Baseline | 4.04 (1.397) | 4.38 (1.719)
  Direct Bilirubin: Week 8: number analyzed (Participants) | 32 | 36
  Direct Bilirubin: Week 8 | -0.06 (1.105) | -0.22 (1.149)
  Direct Bilirubin: Week 16: number analyzed (Participants) | 59 | 61
  Direct Bilirubin: Week 16 | 0.24 (1.088) | -0.28 (1.227)
  Direct Bilirubin: Week 32: number analyzed (Participants) | 18 | 23
  Direct Bilirubin: Week 32 | 0.00 (1.029) | -0.04 (1.147)
  Direct Bilirubin: Week 52: number analyzed (Participants) | 54 | 54
  Direct Bilirubin: Week 52 | 0.28 (1.280) | -0.24 (1.228)

20. Secondary Outcome: Change From Baseline in Gamma Glutamyl Transferase
Description: Change from baseline in gamma glutamyl transferase was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
Units per liter (U/L)
  Baseline | 67.6 (43.02) | 79.4 (45.89)
  Week 8: number analyzed (Participants) | 34 | 37
  Week 8 | -4.8 (13.22) | -5.5 (12.56)
  Week 16: number analyzed (Participants) | 64 | 63
  Week 16 | -4.4 (13.79) | 0.7 (27.43)
  Week 32: number analyzed (Participants) | 19 | 24
  Week 32 | -1.3 (13.39) | -5.3 (23.29)
  Week 52: number analyzed (Participants) | 59 | 58
  Week 52 | -3.2 (22.40) | -6.7 (21.31)

21. Secondary Outcome: Change From Baseline in Creatinine
Description: Change from baseline in creatinine was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micromole/liter (umol/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 67
micromole/liter (umol/L)
  Baseline | 78.1 (14.36) | 78.9 (17.42)
  Week 8: number analyzed (Participants) | 34 | 36
  Week 8 | -2.0 (7.49) | -6.2 (7.49)
  Week 16: number analyzed (Participants) | 64 | 62
  Week 16 | -1.1 (10.72) | -0.3 (12.46)
  Week 32: number analyzed (Participants) | 19 | 24
  Week 32 | 2.2 (10.81) | -1.8 (13.46)
  Week 52: number analyzed (Participants) | 59 | 58
  Week 52 | -1.5 (9.52) | 0.4 (10.00)

22. Secondary Outcome: Change From Baseline in Urea Nitrogen
Description: Change from baseline in urea nitrogen was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
millimoles per liter (mmol/L)
  Baseline | 5.26 (1.402) | 5.08 (1.350)
  Week 8: number analyzed (Participants) | 34 | 37
  Week 8 | -0.30 (0.989) | -0.09 (1.217)
  Week 16: number analyzed (Participants) | 64 | 63
  Week 16 | -0.04 (1.043) | 0.06 (1.278)
  Week 32: number analyzed (Participants) | 19 | 24
  Week 32 | 0.02 (0.955) | -0.25 (1.274)
  Week 52: number analyzed (Participants) | 59 | 68
  Week 52 | -0.06 (1.251) | 0.04 (1.101)

23. Secondary Outcome: Change From Baseline in Urate
Description: Change from baseline in urate was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
umol/L
  Baseline | 360.0 (70.95) | 372.7 (88.25)
  Week 8: number analyzed (Participants) | 34 | 37
  Week 8 | -0.8 (40.76) | -53.6 (40.17)
  Week 16: number analyzed (Participants) | 64 | 62
  Week 16 | 2.8 (40.13) | -37.8 (40.01)
  Week 32: number analyzed (Participants) | 19 | 24
  Week 32 | 16.0 (39.35) | -56.7 (53.18)
  Week 52: number analyzed (Participants) | 59 | 58
  Week 52 | 1.1 (49.36) | -25.8 (54.39)

24. Secondary Outcome: Change From Baseline in Glucose, Cholesterol, Triglycerides, Sodium, Potassium, Chloride and Calcium
Description: Change from baseline in glucose, cholesterol, triglycerides, sodium, potassium, chloride and calcium was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
mmol/L
  Glucose: Baseline | 4.97 (0.772) | 5.15 (0.868)
  Glucose: Week 8: number analyzed (Participants) | 34 | 37
  Glucose: Week 8 | 0.00 (1.028) | -0.46 (0.914)
  Glucose: Week 16: number analyzed (Participants) | 63 | 63
  Glucose: Week 16 | 0.17 (1.153) | -0.04 (1.022)
  Glucose: Week 32: number analyzed (Participants) | 19 | 24
  Glucose: Week 32 | 0.24 (0.911) | -0.12 (0.850)
  Glucose: Week 52: number analyzed (Participants) | 59 | 59
  Glucose: Week 52 | -0.03 (0.883) | -0.28 (1.193)
  Cholesterol: Baseline | 3.653 (0.7454) | 3.705 (0.6676)
  Cholesterol: Week 8: number analyzed (Participants) | 34 | 37
  Cholesterol: Week 8 | -0.182 (0.3808) | -0.238 (0.3807)
  Cholesterol: Week 16: number analyzed (Participants) | 64 | 62
  Cholesterol: Week 16 | -0.065 (0.3994) | -0.190 (0.5139)
  Cholesterol: Week 32: number analyzed (Participants) | 19 | 24
  Cholesterol: Week 32 | 0.060 (0.5185) | -0.059 (0.5364)
  Cholesterol: Week 52: number analyzed (Participants) | 59 | 59
  Cholesterol: Week 52 | -0.065 (0.4308) | -0.093 (0.4243)
  Triglycerides: Baseline | 1.126 (0.4787) | 1.057 (0.4233)
  Triglycerides: Week 8: number analyzed (Participants) | 34 | 37
  Triglycerides: Week 8 | -0.061 (0.5950) | -0.071 (0.3755)
  Triglycerides: Week 16: number analyzed (Participants) | 64 | 63
  Triglycerides: Week 16 | -0.099 (0.3946) | -0.004 (0.4244)
  Triglycerides: Week 32: number analyzed (Participants) | 19 | 24
  Triglycerides: Week 32 | 0.123 (0.4749) | 0.024 (0.5126)
  Triglycerides: Week 52: number analyzed (Participants) | 59 | 58
  Triglycerides: Week 52 | -0.067 (0.5191) | -0.020 (0.4703)
  Sodium: Baseline | 141.2 (1.93) | 140.8 (2.79)
  Sodium: Week 8: number analyzed (Participants) | 34 | 37
  Sodium: Week 8 | -0.5 (2.02) | -0.2 (2.52)
  Sodium: Week 16: number analyzed (Participants) | 64 | 61
  Sodium: Week 16 | -1.1 (2.74) | -0.6 (2.94)
  Sodium: Week 32: number analyzed (Participants) | 19 | 24
  Sodium: Week 32 | -0.7 (3.23) | -0.3 (2.44)
  Sodium: Week 52: number analyzed (Participants) | 59 | 58
  Sodium: Week 52 | -1.1 (2.28) | -1.0 (2.35)
  Potassium: Baseline | 4.364 (0.2695) | 4.391 (0.2885)
  Potassium: Week 8: number analyzed (Participants) | 34 | 37
  Potassium: Week 8 | -0.074 (0.3476) | -0.030 (0.2876)
  Potassium: Week 16: number analyzed (Participants) | 64 | 61
  Potassium: Week 16 | -0.013 (0.3684) | 0.030 (0.3783)
  Potassium: Week 32: number analyzed (Participants) | 19 | 24
  Potassium: Week 32 | -0.011 (0.3957) | -0.033 (0.2599)
  Potassium: Week 52: number analyzed (Participants) | 59 | 58
  Potassium: Week 52 | -0.031 (0.3354) | -0.003 (0.3356)
  Chloride: Baseline | 103.9 (2.19) | 103.3 (3.30)
  Chloride: Week 8: number analyzed (Participants) | 34 | 37
  Chloride: Week 8 | 0.2 (1.71) | 1.3 (2.33)
  Chloride: Week 16: number analyzed (Participants) | 64 | 61
  Chloride: Week 16 | -0.4 (2.88) | 0.3 (2.75)
  Chloride: Week 32: number analyzed (Participants) | 19 | 24
  Chloride: Week 32 | -0.1 (2.37) | 0.3 (2.28)
  Chloride: Week 52: number analyzed (Participants) | 59 | 59
  Chloride: Week 52 | 0.4 (2.44) | 0.4 (2.89)
  Calcium: Baseline | 2.458 (0.0990) | 2.479 (0.1114)
  Calcium: Week 8: number analyzed (Participants) | 34 | 37
  Calcium: Week 8 | -0.006 (0.1096) | -0.062 (0.0999)
  Calcium: Week 16: number analyzed (Participants) | 64 | 63
  Calcium: Week 16 | -0.002 (0.0929) | -0.050 (0.0943)
  Calcium: Week 32: number analyzed (Participants) | 19 | 24
  Calcium: Week 32 | 0.035 (0.0987) | -0.004 (0.1271)
  Calcium: Week 52: number analyzed (Participants) | 59 | 59
  Calcium: Week 52 | -0.021 (0.1083) | -0.035 (0.1093)

25. Secondary Outcome: Change From Baseline in Albumin and Protein
Description: Change from baseline in albumin and protein was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
grams per liter (g/L)
  Albumin: Baseline | 48.64 (3.024) | 49.56 (3.257)
  Albumin: Week 8: number analyzed (Participants) | 34 | 37
  Albumin: Week 8 | -0.74 (2.789) | -1.73 (2.922)
  Albumin: Week 16: number analyzed (Participants) | 64 | 61
  Albumin: Week 16 | 0.61 (2.821) | -0.82 (3.274)
  Albumin: Week 32: number analyzed (Participants) | 19 | 24
  Albumin: Week 32 | 0.79 (3.276) | 0.38 (3.462)
  Albumin: Week 52: number analyzed (Participants) | 59 | 59
  Albumin: Week 52 | -0.08 (3.426) | -0.53 (3.339)
  Protein: Baseline | 75.0 (4.73) | 75.4 (5.24)
  Protein: Week 8: number analyzed (Participants) | 34 | 37
  Protein: Week 8 | -1.5 (4.28) | -3.8 (4.38)
  Protein: Week 16: number analyzed (Participants) | 64 | 63
  Protein: Week 16 | -0.3 (4.62) | -1.9 (4.51)
  Protein: Week 32: number analyzed (Participants) | 19 | 24
  Protein: Week 32 | -0.2 (4.38) | -0.3 (4.60)
  Protein: Week 52: number analyzed (Participants) | 59 | 58
  Protein: Week 52 | -1.8 (5.42) | -2.5 (5.56)

26. Secondary Outcome: Change From Baseline in Alpha Fetoprotein
Description: Change from baseline in alpha fetoprotein was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
micrograms per milliliter (ug/L)
  Baseline | 3.145 (2.0135) | 3.326 (2.2213)
  Week 8: number analyzed (Participants) | 34 | 38
  Week 8 | 0.006 (0.5537) | -0.061 (0.6314)
  Week 16: number analyzed (Participants) | 65 | 65
  Week 16 | 0.055 (0.4373) | 0.160 (0.5667)
  Week 32: number analyzed (Participants) | 18 | 22
  Week 32 | 0.033 (0.3911) | 0.191 (0.5959)
  Week 52: number analyzed (Participants) | 60 | 58
  Week 52 | 0.068 (0.5003) | 0.240 (0.6349)

27. Secondary Outcome: Change From Baseline in Cystatin C
Description: Change from baseline in cystatin C was reported.
Time Frame: Baseline, Week 8, Week 16, Week 32 and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Placebo | Macitentan
Number analyzed (Participants) | 69 | 68
milligrams per liter (mg/L)
  Baseline | 0.742 (0.1047) | 0.718 (0.1190)
  Week 8: number analyzed (Participants) | 33 | 37
  Week 8 | -0.026 (0.0563) | -0.019 (0.0782)
  Week 16: number analyzed (Participants) | 65 | 64
  Week 16 | -0.017 (0.1464) | -0.019 (0.0964)
  Week 32: number analyzed (Participants) | 19 | 24
  Week 32 | -0.038 (0.0659) | -0.021 (0.0701)
  Week 52: number analyzed (Participants) | 59 | 55
  Week 52 | -0.001 (0.0723) | 0.010 (0.0927)

ADVERSE EVENTS:
Time Frame: Up to 56 weeks
Arm/Group | Placebo | Macitentan
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/68
Serious Adverse Events (participants affected / at risk) | 9/69 | 13/68
Other Adverse Events (participants affected / at risk) | 18/69 | 15/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=69) | Macitentan (N=68)
Arrhythmia Supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Congestive Hepatopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr Virus Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Heart Rate Increased (Investigations) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 1 (1)
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1)
Polydipsia Psychogenic (Psychiatric disorders) | 0 (0) | 1 (1)
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Medical Device Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=69) | Macitentan (N=68)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (6) | 1 (1)
Headache (Nervous system disorders) | 6 (10) | 7 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT03153137/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT03153137/SAP_001.pdf